CLINICAL TRIAL: NCT02393638
Title: ERCP Mechanical Simulator (EMS) Practice for Training Endoscopic Sphincterotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 201403004RIND
Record Dates: First submitted 2015-02-10; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Endoscopic Sphincterotomy
Keywords: Endoscopic Sphincterotomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): Simulation and lecture
  Interventions: Other: Simulation and lecture
- control group (Active Comparator): Lecture only
  Interventions: Other: Lecture

INTERVENTIONS:
Other: Simulation and lecture — Endoscopic sphincterotomy on simulator and lecture
  Arms: study group
Other: Lecture — Lecture
  Arms: control group

SUMMARY:
This randomized-controlled study aims to evaluate the effectiveness of using ERCP mechanical simulator for training endoscopic sphincterotomy.

DETAILED DESCRIPTION:
Usual clinical ERCP training is supervised hands-on practice and the number of procedures is used as a surrogate for trainees' experience. At least 180 cases are required to achieve ERCP competence. A major limitation is lack of suitable patients. Alternative supplemental training includes simulator practice using computer simulators, live animal models, and ex-vivo porcine organ. Our previous study has showed that the mechanical simulator training improves trainees' clinical performance in terms of success of deep CBD cannulation. In this study, we aim to evaluate the usefulness of ERCP mechanical simulator for training endoscopic sphincterotomy.

ELIGIBILITY:
Inclusion Criteria:

* GI trainees who met the minimum endoscopy training experience

Exclusion Criteria:

* GI trainees with no endoscopy experience

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
proportion of endoscopic sphincterotomy successfully performed by trainees | 1year

SECONDARY OUTCOMES:
Improvement in overall performance as measured by sphincterotomy score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: W C Liao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Gastroenterology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Liao WC, Leung JW, Wang HP, Chang WH, Chu CH, Lin JT, Wilson RE, Lim BS, Leung FW. Coached practice using ERCP mechanical simulator improves trainees' ERCP performance: a randomized controlled trial. Endoscopy. 2013 Oct;45(10):799-805. doi: 10.1055/s-0033-1344224. Epub 2013 Jul 29. PMID 23897401